CLINICAL TRIAL: NCT03635112
Title: A Phase 2 Multi-Center, Randomized, Double-Blind, Placebo˗Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Induction Therapy With 2 Doses of TD-1473 in Subjects With Moderately-to-Severely Active Crohn's Disease
Brief Title: Efficacy and Safety of TD-1473 in Crohn's Disease
Acronym: DIONE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated by the sponsor on 16 November 2021 after a planned review by the Independent Data Monitoring Committee.
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0173; 2018-001272-37 (EudraCT Number)
Record Dates: First submitted 2018-07-31; First posted 2018-08-17 (Actual); Results first posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-02

CONDITIONS: Crohn's Disease
Keywords: TD-1473; Janus kinase inhibitor; JAK inhibitor; Inflammatory Bowel Disease; IBD; Crohn's Disease; Intestinal restriction
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — izencitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Active Treatment TD-1473 with Dose A (Active Comparator): 1 oral Dose A daily of TD-1473 for 12 weeks in subjects with moderately to-severely active CD.
  Subjects who complete Induction will continue to receive TD-1473 at Dose A in the Active Treatment Arm for up to 48 additional weeks.
  Interventions: Drug: TD-1473
- Active Treatment TD-1473 with Dose B (Active Comparator): 1 oral Dose B daily of TD-1473 for 12 weeks in subjects with moderately to-severely active CD.
  Subjects who complete Induction will continue to receive TD-1473 at Dose B in the Active Treatment Arm for up to 48 additional weeks.
  Interventions: Drug: TD-1473
- Placebo (Placebo Comparator): 1 oral dose daily of placebo for 12 weeks in subjects with moderately to-severely active CD.
  Subjects who complete Induction will receive TD-1473 at Dose A in the Active Treatment Arm for up to 48 additional weeks.
  Interventions: Drug: Placebo; Drug: TD-1473

INTERVENTIONS:
Drug: Placebo — Placebo will be taken daily by mouth (orally) for up to 12 weeks in the morning before eating.
  Arms: Placebo
Drug: TD-1473 — TD-1473, at Dose A or Dose B depending upon arm, will be taken daily by mouth (orally) for up to 12 weeks in the morning before eating. An additional 48 weeks either at Dose A or Dose B, depending on arm, may be administered if subjects finish the 12 week induction period.

SUMMARY:
A Phase 2 study to evaluate the efficacy, safety and tolerability of TD-1473 in subjects with moderately-to-severely active Crohn's Disease with up to 48 weeks of treatment.

DETAILED DESCRIPTION:
A Phase 2 multi-center, randomized, double blind, placebo-controlled, parallel-group study to evaluate the efficacy and safety of 12 weeks of induction therapy with TD˗1473 in subjects with moderately-to-severely active Crohn's Disease. This study includes 3 phases: Screening, Induction, and Active Treatment Extension (ATE). The Induction phase of the study is a randomized, double blind, placebo controlled, parallel group study evaluating 2 oral dose levels of TD-1473 compared to placebo for 12 weeks in subjects with moderately to-severely active CD. Subjects who complete Induction will continue to receive TD-1473 in the ATE, for up to 48 additional weeks.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age at screening
* Males and females with clinical evidence of Crohn's disease for at least 3 months duration at screening
* Moderately-to-severely active Crohn's Disease at baseline, as defined by a Crohn's Disease Activity Index (CDAI) score of 220-450 inclusive
* SES-CD score of ≥ 3 with ulceration (corresponding to a score of 1) in at least 1 of the 5 ileocolonic segments on the Ulcerated Surface subscore of the SES-CD]
* Is corticosteroid-dependent or has demonstrated inadequate response, or intolerance to conventional therapy (aminosalicylates, corticosteroids and immunomodulators such as azathioprine, 6-mercaptopurine, or methotrexate) or biologics (e.g., anti-TNF therapy, anti-IL-12/23 (anti-interleukin), anti-integrin).
* Additional inclusion criteria apply

Exclusion Criteria:

* Is currently receiving biologic (anti-TNF, anti-integrin, or anti-IL12/23) therapy
* Has a current bacterial, parasitic, fungal, or viral infection
* Has clinically significant abnormalities in laboratory evaluations
* Prior exposure or potential exposure to a JAK inhibitor that was stopped due to intolerance or lack of efficacy
* Subject has participated in another clinical trial of an investigational drug (or medical device) within 30 days prior to Screening or 5x the half-life of the investigational drug, whichever is longer, or is currently participating in another trial of an investigational drug (or medical device)
* Subject has failed ≥ 3 biologic agents of 3 different mechanisms of action (i.e., anti-TNF, anti-integrin, and anti-IL12/23)
* Additional exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (152):
- United States (42):
  - Theravance Biopharma Investigational Site, Birmingham, Alabama
  - Theravance Biopharma Investigational Site, Mobile, Alabama
  - Theravance Biopharma Investigational Site, Scottsdale, Arizona
  - Theravance Biopharma Investigational Site, La Jolla, California
  - Theravance Biopharma Investigational Site, Los Angeles, California
  - Theravance Biopharma Investigational Site, Oakland, California
  - Theravance Biopharma Investigational Site, Santa Monica, California
  - Theravance Biopharma Investigational Site, Aventura, Florida
  - Theravance Biopharma Investigational Site, Clearwater, Florida
  - Theravance Biopharma Investigational Site, Hialeah, Florida
  - Theravance Biopharma Investigational Site, Hollywood, Florida
  - Theravance Biopharma Investigational Site, Largo, Florida
  - Theravance Biopharma Investigational Site, Miami, Florida
  - Theravance Biopharma Investigational Site, New Port Richey, Florida
  - Theravance Biopharma Investigational Site, St. Petersburg, Florida
  - Theravance Biopharma Investigational Site, Tampa, Florida
  - Theravance Biopharma Investigational Site, New Lenox, Illinois
  - Theravance Biopharma Investigational Site, Kansas City, Kansas
  - Theravance Biopharma Investigational Site, Louisville, Kentucky
  - Theravance Biopharma Investigational Site, Rockville, Maryland
  - Theravance Biopharma Investigational Site, Brockton, Massachusetts
  - Theravance Biopharma Investigational Site, Wyoming, Michigan
  - Theravance Biopharma Investigational Site, St Louis, Missouri
  - Theravance Biopharma Investigational Site, Las Vegas, Nevada
  - Theravance Biopharma Investigational Site, Utica, New York
  - Theravance Biopharma Investigational Site, Gastonia, North Carolina
  - Theravance Biopharma Investigational Site, Greenville, North Carolina
  - PMG Research of Salisbury, Salisbury, North Carolina
  - Theravance Biopharma Investigational Site, Tulsa, Oklahoma
  - Theravance Biopharma Investigational Site, Pittsburgh, Pennsylvania
  - Theravance Biopharma Investigational Site, Uniontown, Pennsylvania
  - Theravance Biopharma Investigational Site, Orangeburg, South Carolina
  - Theravance Biopharma Investigational Site, Rock Hill, South Carolina
  - Theravance Biopharma Investigational Site, Boerne, Texas
  - Theravance Biopharma Investigational Site, El Paso, Texas
  - Theravance Biopharma Investigational Site, Garland, Texas
  - Theravance Biopharma Investigational Site, Harlingen, Texas
  - Theravance Biopharma Investigational Site, Houston, Texas
  - Theravance Biopharma Investigational Site, San Antonio, Texas
  - Theravance Biopharma Investigational Site, Southlake, Texas
  - Theravance Biopharma Investigational Site, Spring, Texas
  - Theravance Biopharma Investigational Site, Lansdowne Town Center, Virginia
- Australia (3):
  - Theravance Biopharma Investigational Site, Bankstown, New South Wales
  - Theravance Biopharma Investigational Site, Elizabeth Vale, South Australia
  - Theravance Biopharma Investigational Site, Perth, Western Australia
- Austria (3):
  - Theravance Biopharma Investigational Site, Klagenfurt, Carinthia
  - Theravance Biopharma Investigational Site, Innsbruck, Tyrol
  - Theravance Biopharma Investigational Site, Vienna, Vienna
- Bulgaria (7):
  - Theravance Biopharma Investigational Site, Sofia, Sofia
  - Theravance Biopharma Investigational Site, Targovishte, Targovishte
  - Theravance Biopharma Investigational Site, Dobrich
  - Theravance Biopharma Investigational Site, Plovdiv
  - Theravance Biopharma Investigational Site, Sliven
  - Theravance Biopharma Investigational Site, Stara Zagora
  - Theravance Biopharma Investigational Site, Veliko Tarnovo
- Croatia (4):
  - Theravance Biopharma Investigational Site, Osijek, County of Osijek-Baranja
  - Theravance Biopharma Investigational Site, Rijeka
  - Theravance Biopharma Investigational Site, Split
  - Theravance Biopharma Investigational Site, Zagreb
- France (8):
  - Theravance Biopharma Investigational Site, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Theravance Biopharma Investigational Site, Saint-Etienne, Auvergne
  - Theravance Biopharma Investigational Site, Reims, Champagne-ardenne
  - Theravance Biopharma Investigational Site, Toulouse, Midi-pyrenees
  - Theravance Biopharma Investigational Site, Nice, Provence-Alpes-Côte d'Azur Region
  - Theravance Biopharma Investigational Site, Clichy
  - Theravance Biopharma Investigational Site, Vandœuvre-lès-Nancy
  - Theravance Biopharma Investigational Site, Colombes, Île-de-France Region
- Theravance Biopharma Investigational Site, Tbilisi, Georgia
- Germany (5):
  - Theravance Biopharma Investigational Site, München, Bavaria
  - Theravance Biopharma Investigational Site, Hanover, Lower Saxony
  - Theravance Biopharma Investigational Site, Kiel, Schleswig-Holstein
  - Theravance Biopharma Investigational Site, Berlin
  - Theravance Biopharma Investigational Site, Hamburg
- Greece (2):
  - Theravance Biopharma Investigational Site, Athens, Attica
  - Theravance Biopharma Investigational Site, Heraklion, Crete
- Hungary (4):
  - Theravance Biopharma Investigational Site, Baja, Bács-Kiskun county
  - Theravance Biopharma Investigational Site, Debrecen, Hajdú-Bihar
  - Theravance Biopharma Investigational Site, Gyöngyös, Heves County
  - Theravance Biopharma Investigational Site, Budapest
- Israel (9):
  - Theravance Biopharma Investigational Site, Be’er Ya‘aqov, Rehoboth
  - Theravance Biopharma Investigational Site, Rehovot, Rehoboth
  - Theravance Biopharma Investigational Site, Kfar Saba, Sharon
  - Theravance Biopharma Investigational Site, Haifa
  - Theravance Biopharma Investigational Site, Holon
  - Theravance Biopharma Investigational Site, Jerusalem
  - Theravance Biopharma Investigational Site, Nahariya
  - Theravance Biopharma Investigational Site, Petah Tikva
  - Theravance Biopharma Investigational Site, Tel Aviv
- New Zealand (2):
  - Theravance Biopharma Investigational Site, Hamilton, Waikato Region
  - Theravance Biopharma Investigational Site, Lower Hutt, Wellington Region
- Poland (10):
  - Theravance Biopharma Investigational Site, Poznan, Greater Poland Voivodeship
  - Theravance Biopharma Investigational Site, Włocławek, Kuyavian-Pomeranian Voivodeship
  - Theravance Biopharma Investigational Site, Krakow, Lesser Poland Voivodeship
  - Theravance Biopharma Investigational Site, Wroclaw, Lower Silesian Voivodeship
  - Theravance Biopharma Investigational Site, Warsaw, Masovian Voivodeship
  - Theravance Biopharma Investigational Site, Rzeszów, Podkarpackie Voivodeship
  - Theravance Biopharma Investigational Site, Sopot, Pomeranian Voivodeship
  - Theravance Biopharma Investigational Site, Tychy, Silesian Voivodeship
  - Theravance Biopharma Investigational Site, Szczecin, Zachodnio-Pomorskie
  - Theravance Biopharma Investigational Site, Lodz, Łódź Voivodeship
- Portugal (7):
  - Theravance Biopharma Investigational Site, Braga
  - Theravance Biopharma Investigational Site, Guimarães
  - Theravance Biopharma Investigational Site, Leiria
  - Theravance Biopharma Investigational Site, Lisbon
  - Theravance Biopharma Investigational Site, Santa Maria da Feira
  - Theravance Biopharma Investigational Site, Setúbal
  - Theravance Biopharma Investigational Site, Vila Nova de Gaia
- Romania (6):
  - Theravance Biopharma Investigational Site, Oradea, Bihor County
  - Theravance Biopharma Investigational Site, Bucharest, București
  - Theravance Biopharma Investigational Site, Cluj-Napoca, Cluj
  - Theravance Biopharma Investigational Site, Timișoara, Timiș County
  - Theravance Biopharma Investigational Site, Bucharest
  - Theravance Biopharma Investigational Site, Cluj-Napoca
- Russia (6):
  - Theravance Biopharma Investigational Site, Moscow, Moscow City
  - Theravance Biopharma Investigational Site, Rostov-on-Don, Rostov Oblast
  - Theravance Biopharma Investigational Site, Samara, Samara Oblast
  - Theravance Biopharma Investigational Site, Novosibirsk
  - Theravance Biopharma Investigational Site, Saint Petersburg
  - Theravance Biopharma Investigational Site, Saratov
- Serbia (5):
  - Theravance Biopharma Investigational Site, Belgrade
  - Theravance Biopharma Investigational Site, Kragujevac
  - Theravance Biopharma Investigational Site, Niš
  - Theravance Biopharma Investigational Site, Subotica
  - Theravance Biopharma Investigational Site, Zrenjanin
- South Africa (3):
  - Theravance Biopharma Investigational Site, Johannesburg, Gauteng
  - Theravance Biopharma Investigational Site, Lenasia, Gauteng
  - Theravance Biopharma Investigational Site, Claremont, Western Cape
- South Korea (6):
  - Theravance Biopharma Investigational Site, Wŏnju, Gangwon-do
  - Theravance Biopharma Investigational Site, Guri-si, Gyeonggi-do
  - Theravance Biopharma Investigational Site, Seongnam-si, Gyeonggi-do
  - Theravance Biopharma Investigational Site, Busan
  - Theravance Biopharma Investigational Site, Daegu
  - Theravance Biopharma Investigational Site, Seoul
- Spain (5):
  - Theravance Biopharma Investigational Site, Las Palmas de Gran Canaria, Las Palmas
  - Theravance Biopharma Investigational Site, Barcelona
  - Theravance Biopharma Investigational Site, Huelva
  - Theravance Biopharma Investigational Site, Madrid
  - Theravance Biopharma Investigational Site, Valencia
- Ukraine (11):
  - Theravance Biopharma Investigational Site, Kiev, KIEV CITY
  - Theravance Biopharma Investigational Site, Kyiv, KIEV CITY
  - Theravance Biopharma Investigational Site, Kyiv, Kyiv City
  - Theravance Biopharma Investigational Site, Kremenchuk, Poltava Oblast
  - Theravance Biopharma Investigational Site, Uzhhorod, Transcarpathian
  - Theravance Biopharma Investigational Site, Uzhhorod, Zakarpattia Oblast
  - Theravance Biopharma Investigational Site, Chernivtsi
  - Theravance Biopharma Investigational Site, Kharkiv
  - Theravance Biopharma Investigational Site, Lviv
  - Theravance Biopharma Investigational Site, Vinnytsia
  - Theravance Biopharma Investigational Site, Zaporizhzhya
- United Kingdom (3):
  - Theravance Biopharma Investigational Site, Blackpool, England
  - Theravance Biopharma Investigational Site, London, England
  - Theravance Biopharma Investigational Site, Glasgow, Scotland

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 167 participants were randomized, of which 159 were eligible for analysis at sites in Australia, Asia/Pacific, Israel, Russia, the United States and South Africa between 19 November 2018 and 30 December 2021.
Groups:
- Placebo: Participants were randomized to receive once-daily oral administrations of placebo for 12 weeks during the Induction Period. Participants who completed the Induction Period received once-daily oral administrations of TD-1473 80 mg in the Active Treatment Extension period for up to 48 additional weeks.
- TD-1473 80 mg: Participants were randomized to receive once-daily oral administrations of TD-1473 80 mg for 12 weeks during the Induction Period. Participants who completed the Induction Period received once-daily oral administrations of TD-1473 80 mg in the Active Treatment Extension period for up to 48 additional weeks.
- TD-1473 200 mg: Participants were randomized to receive once-daily oral administrations of TD-1473 200 mg for 12 weeks during the Induction Period. Participants who completed the Induction Period received once-daily oral administrations of TD-1473 200 mg in the Active Treatment Extension period for up to 48 additional weeks.
Period: Overall Study
Arm/Group | Placebo | TD-1473 80 mg | TD-1473 200 mg
Started | 38 | 58 | 63
Completed Week 12 Visit | 33 | 48 | 49
Switched From Placebo to TD-1473 80 mg | 33 | 0 | 0
Completed | 12 | 16 | 13
Not Completed | 26 | 42 | 50
Not completed — Adverse Event | 5 | 9 | 14
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Physician Decision | 5 | 7 | 5
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 11 | 17 | 21
Not completed — Withdrawal by Subject | 4 | 9 | 7
Not completed — Miscellaneous | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Analysis Set: Comprised all randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TD-1473 80 mg | TD-1473 200 mg | Total
Number analyzed (Participants) | 38 | 58 | 63 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (14.85) | 37.1 (12.45) | 40.0 (13.64) | 38.8 (13.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 28 | 31 | 77
  Male | 20 | 30 | 32 | 82
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 3
  Not Hispanic or Latino | 36 | 57 | 60 | 153
  Unknown | 0 | 0 | 2 | 2
  Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Crohn's Disease Activity Index (CDAI) Score
Description: The CDAI score was generated using regression coefficients for eight different predictors of disease activity: severity of abdominal pain, general well-being, very soft/liquid stool frequency, extra-intestinal symptoms, need for antidiarrheal drugs, presence of an abdominal mass, body weight and hematocrit. Participants reported information regarding symptoms using a diary. The subscores of abdominal pain (0-3), general well-being (0-4), and number of very soft or liquid stools were then summed over the 7 days prior to each visit. Additionally, the remaining predictors were also noted and weighted to create the total CDAI score which ranged from 0-600 with a higher score indicating a worse outcome.
  Benchmarks for disease activity as measured by the CDAI were: <150, clinical remission; 150 to 219, mildly active disease; 220-450, moderately active disease; and >450, very severe disease.
Time Frame: Baseline to Week 12
Population: Modified Intent-to-Treat Analysis Set: Comprised all randomized evaluable participants who received at least 1 dose of study drug, had at least one postbaseline CDAI score and had non-missing values at both baseline and postbaseline visit.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TD-1473 80 mg | TD-1473 200 mg
Number analyzed (Participants) | 33 | 47 | 50
score on a scale | -104.86 (15.496) | -105.62 (12.713) | -117.99 (12.423)
Statistical Analysis 1: Comparison: Placebo vs TD-1473 80 mg; Test type: Superiority; p = 0.970, Mixed Model Repeated Measures Analysis; Least Square Mean Difference = -0.76, 95% CI 2-sided [-40.62 to 39.11]
Statistical Analysis 2: Comparison: Placebo vs TD-1473 200 mg; Test type: Superiority; p = 0.510, Mixed Model Repeated Measures Analysis; Least Square Mean Difference = -13.13, 95% CI 2-sided [-52.46 to 26.19]

2. Secondary Outcome: Number of Participants Who Demonstrated a Clinical Response as Measured by CDAI
Description: The CDAI score was generated using regression coefficients for eight different predictors of disease activity: severity of abdominal pain, general well-being, very soft/liquid stool frequency, extra-intestinal symptoms, need for antidiarrheal drugs, presence of an abdominal mass, body weight and hematocrit. Participants reported information regarding symptoms using a diary. The subscores of abdominal pain (0-3), general well-being (0-4), and number of very soft or liquid stools were then summed over the 7 days prior to each visit. Additionally, the remaining predictors were also noted and weighted to create the total CDAI score which ranged from 0-600 with a higher score indicating a worse outcome.
  Benchmarks for disease activity as measured by the CDAI were: <150, clinical remission; 150 to 219, mildly active disease; 220-450, moderately active disease; and >450, very severe disease.
  Clinical response was defined as a reduction from baseline of ≥100 points or CDAI <150
Time Frame: Week 12
Population: Modified Intent-to-Treat Analysis Set: Comprised all randomized evaluable participants who received at least 1 dose of study drug and had at least one postbaseline CDAI score.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TD-1473 80 mg | TD-1473 200 mg
Number analyzed (Participants) | 35 | 54 | 56
Participants | 19 | 28 | 34
Statistical Analysis 1: Comparison: Placebo vs TD-1473 80 mg; Test type: Superiority; p = 0.5102, Cochran-Mantel-Haenszel Chi-square Test; Difference in Proportion = -0.07, 95% CI 2-sided [-0.277 to 0.135]
Statistical Analysis 2: Comparison: Placebo vs TD-1473 200 mg; Test type: Superiority; p = 0.8591, Cochran-Mantel-Haenszel Chi-square Test; Difference in Proportion = 0.02, 95% CI 2-sided [-0.181 to 0.218]

3. Secondary Outcome: Number of Participants Who Demonstrated CDAI Clinical Remission
Description: The CDAI score was generated using regression coefficients for eight different predictors of disease activity: severity of abdominal pain, general well-being, very soft/liquid stool frequency, extra-intestinal symptoms, need for antidiarrheal drugs, presence of an abdominal mass, body weight and hematocrit. Participants reported information regarding symptoms using a diary. The subscores of abdominal pain (0-3), general well-being (0-4), and number of very soft or liquid stools were then summed over the 7 days prior to each visit. Additionally, the remaining predictors were also noted and weighted to create the total CDAI score which ranged from 0-600 with a higher score indicating a worse outcome.
  Benchmarks for disease activity as measured by the CDAI were: <150, clinical remission; 150 to 219, mildly active disease; 220-450, moderately active disease; and >450, very severe disease.
  CDAI clinical remission was defined as a CDAI score less than 150 at Week 12.
Time Frame: Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TD-1473 80 mg | TD-1473 200 mg
Number analyzed (Participants) | 35 | 54 | 56
Participants | 13 | 13 | 22
Statistical Analysis 1: Comparison: Placebo vs TD-1473 80 mg; Test type: Superiority; p = 0.1805, Cochran-Mantel-Haenszel Chi-square Test; Difference in Proportion = -0.13, 95% CI 2-sided [-0.322 to 0.061]
Statistical Analysis 2: Comparison: Placebo vs TD-1473 200 mg; Test type: Superiority; p = 0.9215, Cochran-Mantel-Haenszel Chi-square Test; Difference in Proportion = -0.01, 95% CI 2-sided [-0.204 to 0.184]

4. Secondary Outcome: Change From Baseline in Simple Endoscopic Score for Crohn's Disease (SES-CD) at Week 12
Description: The SES-CD incorporated 4 descriptors: the ulcer size, the proportion of surface covered by ulcer, the proportion of surface covered by other lesions, and the presence of stenosis. Each descriptor was scored in 5 segments (ileum, right colon, transverse colon, left colon, and rectum). The total score ranged from 0 to 56, with higher scores indicating a worse outcome.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TD-1473 80 mg | TD-1473 200 mg
Number analyzed (Participants) | 20 | 35 | 37
score on a scale | -1.9 (1.27) | -0.2 (0.96) | -1.9 (0.95)
Statistical Analysis 1: Comparison: Placebo vs TD-1473 80 mg; Test type: Superiority; p = 0.316, ANCOVA; Least Square Mean Difference = 1.6, 95% CI 2-sided [-1.6 to 4.8]
Statistical Analysis 2: Comparison: Placebo vs TD-1473 200 mg; Test type: Superiority; p = 0.988, ANCOVA; Least Square Mean Difference = -0.0, 95% CI 2-sided [-3.2 to 3.2]

5. Secondary Outcome: Number of Participants With Endoscopic Response at Week 12
Description: Endoscopic Response was defined as a reduction of SES-CD score or Endoscopic Remission (defined as SES-CD ≤ 2) at Week 12.
Time Frame: Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TD-1473 80 mg | TD-1473 200 mg
Number analyzed (Participants) | 31 | 53 | 54
Participants | 6 | 5 | 15
Statistical Analysis 1: Comparison: Placebo vs TD-1473 80 mg; Test type: Superiority; p = 0.1828, Cochran-Mantel-Haenszel Chi-square Test; Difference in Proportion = -0.11, 95% CI 2-sided [-0.270 to 0.059]
Statistical Analysis 2: Comparison: Placebo vs TD-1473 200 mg; Test type: Superiority; p = 0.5785, Cochran-Mantel-Haenszel Chi-square Test; Difference in Proportion = 0.06, 95% CI 2-sided [-0.133 to 0.244]

6. Secondary Outcome: Number of Participants With Stool Frequency and Abdominal Pain (SFAP) Clinical Remission
Description: SFAP clinical remission was defined as an abdominal pain score ≤1 (on a scale of 0-3 with 0 representing 'no pain' and 3 representing 'severe pain'), stool frequency ≤2.8, and both not worse than baseline at Week 12.
Time Frame: Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TD-1473 80 mg | TD-1473 200 mg
Number analyzed (Participants) | 35 | 54 | 56
Participants | 6 | 6 | 10
Statistical Analysis 1: Comparison: Placebo vs TD-1473 80 mg; Test type: Superiority; p = 0.3776, Cochran-Mantel-Haenszel Chi-square Test; Difference in Proportion = -0.07, 95% CI 2-sided [-0.225 to 0.095]
Statistical Analysis 2: Comparison: Placebo vs TD-1473 200 mg; Test type: Superiority; p = 0.6063, Cochran-Mantel-Haenszel Chi-square Test; Difference in Proportion = -0.04, 95% CI 2-sided [-0.189 to 0.111]

ADVERSE EVENTS:
Time Frame: From Day 1 up to 28 days after the last dose (up to 64 weeks)
Description: The safety analysis set comprised all participants who received at least 1 dose of study drug.
Groups:
- TD-1473 80mg Post-Placebo: Participants who were treated with placebo in Induction Period and switched to TD-1473 80mg in Active Treatment Extension period.
Arm/Group | Placebo | TD-1473 80 mg | TD-1473 80mg Post-Placebo | TD-1473 200 mg
All-Cause Mortality (participants affected / at risk) | 1/38 | 0/58 | 0/33 | 0/63
Serious Adverse Events (participants affected / at risk) | 3/38 | 9/58 | 3/33 | 10/63
Other Adverse Events (participants affected / at risk) | 11/38 | 23/58 | 7/33 | 22/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=38) | TD-1473 80 mg (N=58) | TD-1473 80mg Post-Placebo (N=33) | TD-1473 200 mg (N=63)
Crohn's Disease (Gastrointestinal disorders) | 0 | 6 | 1 | 8
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intussusception (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Granuloma (General disorders) | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=38) | TD-1473 80 mg (N=58) | TD-1473 80mg Post-Placebo (N=33) | TD-1473 200 mg (N=63)
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 4
Anaemia (Blood and lymphatic system disorders) | 0 | 4 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 3
Crohn's disease (Gastrointestinal disorders) | 3 | 8 | 2 | 7
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 0 | 1
Headache (Nervous system disorders) | 3 | 3 | 1 | 5
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 5
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 4 | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 1 | 0 | 4
Urinary tract infection (Infections and infestations) | 1 | 4 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 1

LIMITATIONS AND CAVEATS:
The study was terminated by the sponsor on 16 November 2021 after a planned review by the Independent Data Monitoring Committee.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/12/NCT03635112/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-27): https://cdn.clinicaltrials.gov/large-docs/12/NCT03635112/SAP_001.pdf